CLINICAL TRIAL: NCT00121849
Title: A Phase 1, Open-Label Study to Evaluate the Safety, Tolerability, and Immunogenicity of the Leish-111f + MPL-SE Vaccine in Montenegro Skin Test-Positive Healthy Adults
Brief Title: Safety Study to Evaluate the Leish-111f + MPL-SE Vaccine in the Prevention of Cutaneous Leishmaniasis in Healthy Subjects Previously Exposed to the Leishmania Parasite
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Access to Advanced Health Institute (AAHI) (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IDRI-LCVPX-105
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 2006-05

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Leishmaniasis,; Subunit Vaccine,; Prevention,; T cell
MeSH Terms: conditions — Leishmaniasis, Cutaneous; Leishmaniasis

INTERVENTIONS:
Biological: Leish-111f + MPL-SE vaccine

SUMMARY:
This study will evaluate the safety of the Leish-111f + MPL-SE vaccine in adult subjects with a previous exposure to the Leishmania parasite (but without current or past history of leishmaniasis).

DETAILED DESCRIPTION:
Cutaneous leishmaniasis is a disfiguring disease that can progress to mucosal leishmaniasis, a more serious and possibly fatal form of Leishmania disease. All available medical therapies require weeks of treatment and cause significant toxicity. It appears that Leishmania infections can be eliminated or prevented by T helper 1 immune responses. These findings argue that a vaccine that generates a T helper 1 response against the parasite will prevent the infection and disease. This is a phase 1, open-label study to evaluate the safety, tolerability and immunogenicity in Montenegro skin test (MST)-positive healthy adults of an investigational vaccine being developed for the prophylaxis of cutaneous leishmaniasis. The vaccine, identified as Leish-111f + MPL-SE, consists of a recombinant three-antigen Leishmania polyprotein (Leish-111f, 10 μg) together with the adjuvant MPL-SE (25 μg). The vaccine will be given to each study subject three times at 4 week intervals.

ELIGIBILITY:
Inclusion Criteria:

* Must have positive Montenegro skin test (reaction >5 mm)
* Must be in good general health with normal lab values
* Negative for HIV, hepatitis B and C

Exclusion Criteria:

* History of leishmaniasis or exposure to Leishmania vaccine or MPL-SE.
* Pregnant or nursing female

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2005-08; Study Completion 2006-02

PRIMARY OUTCOMES:
Adverse events
Dose-limiting toxicities: hematology and serum chemistries at Screening and Days 7, 35, 63, and 84

SECONDARY OUTCOMES:
IgG and T-cell responses to the Leish-111f protein: immunological evaluations at Days 0, 84, and 168
Skin test reactivity to the Leish-111f protein at Days 0, 84, and 168

CONTACTS AND LOCATIONS:
Overall Officials: Iván D Vélez Bernal, MD, PhD, Principal Investigator — PECET, Medellin, Colombia
Locations (1):
- Programa de Estudio y Control de Enfermedades Tropicales (PECET), Medellín, Colombia